CLINICAL TRIAL: NCT06796361
Title: Role of the Serotonin 2A Receptor in Psilocybin-induced Altered States of Consciousness (PDR-Study)
Brief Title: Role of the Serotonin 2A Receptor in Psilocybin-induced Altered States of Consciousness
Acronym: PDR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BASEC 2024-01503; BASEC 2024-01503 (Other: EKNZ)
Record Dates: First submitted 2025-01-13; First posted 2025-01-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: Hallucinogens; Physiological Effects of Drugs; Psychotropic Drugs; Serotonin Antagonists; Serotonin Agents; Neurotransmitter Agents; Molecular Mechanisms of Pharmacological Action; Serotonin Receptor Agonists; Psilocybin
MeSH Terms: interventions — Ketanserin; Psilocybin

STUDY DESIGN:
Intervention Model Description: 6-period random order, placebo-controlled, double-blind cross-over study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 40mg Psilocybin plus 40mg Ketanserin (Experimental): 40mg Ketanserin oral followed by 40mg Psilocybin oral one hour later
  Interventions: Drug: Ketanserin 40mg plus Psilocybin 40mg
- 40mg Psilocybin (Experimental): 40mg Psilocybin oral
  Interventions: Drug: 40mg Psilocybin
- 20mg Psilocybin (Experimental): 20mg Psilocybin oral
  Interventions: Drug: 20mg Psilocybin
- 10mg Psilocybin (Experimental): 10mg Psilocybin oral
  Interventions: Drug: 10mg Psilocybin
- 5mg Psilocybin (Experimental): 5mg Psilocybin oral
  Interventions: Drug: 5mg Psilocybin
- Placebo (Placebo Comparator): Placebo followed by Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketanserin 40mg plus Psilocybin 40mg — 40mg Ketanserin oral will be administered followed by 40mg Psilocybin.
  Arms: 40mg Psilocybin plus 40mg Ketanserin
Drug: 40mg Psilocybin — Placebo oral followed by 40mg Psilocybin one hour later.
  Arms: 40mg Psilocybin
Drug: 20mg Psilocybin — Placebo oral followed by 20mg Psilocybin one hour later.
  Arms: 20mg Psilocybin
Drug: 10mg Psilocybin — Placebo oral followed by 10mg Psilocybin oral one hour later.
  Arms: 10mg Psilocybin
Drug: 5mg Psilocybin — Placebo oral followed by 5mg Psilocybin one hour later
  Arms: 5mg Psilocybin
Other: Placebo — Oral Placebo followed by oral Placebo one hour later
  Arms: Placebo

SUMMARY:
Psilocybin (active compound of "magic mushrooms") is a prototypical psychedelic substance that acts via agonism on serotonin (5-HT) 2A receptors. Psilocybin is rapidly metabolized into its active metabolite psilocin. Psilocybin is currently under investigation as potential treatment for various neuropsychiatric disorders. Psilocybin is also widely used for recreational purposes and as research tool in neuroscience. Besides its current clinical development, a clear characterization of the dose-response relationship of psilocybin is lacking. With the present study the investigators aim to close this knowledge gap by administering low (5mg) to high (40mg) single doses of psilocybin to healthy participants. Besides its agonism on 5-HT2A receptors, psilocin also binds to other receptors and inhibits serotonin transporters (SERT). To this data only few studies have investigated these effects and never at a high dose.

DETAILED DESCRIPTION:
Psilocybin is widely used for recreational and spiritual purposes. Additionally Psilocybin is currently reused in experimental studies with healthy subjects and in studies investigating its effects on patients suffering from anxiety, depression, addiction personality disorders and other pathological conditions.

The present PDR-study will characterize the subjective effects of different doses of psilocybin using modern psychometric instruments, explore the relationship between the plasma-concentration of psilocybin and its subjective effects, and examine the contribution of the 5-HT2A receptor in the psilocybin-induced alterations of consciousness in a mechanistic study in healthy subjects.

Participants will recieve doses of 5, 10, 20, and 40 mg psilocybin, 40 mg of psilocybin with pretreatment of 40 mg ketanserin, and placebo (control for psilocybin). Placebo pretreatment (control for ketanserin) will be used for all psilocybin administrations without ketanserin. Administrations will be separated by at least 10 days and are in random and counter-balanced order.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 75 years.
2. Sufficient understanding of the German language.
3. Understanding the procedures and the risks that are associated with the study.
4. Participants must be willing to adhere to the protocol and sign the consent form.
5. Participants must be willing to refrain from taking illicit psychoactive substances during the study (not including cannabis).
6. Participants must be willing not to drive a traffic vehicle or to operate machines within 48 h after substance administration.
7. Women of childbearing potential must be willing to use effective birth-control throughout study participation

Exclusion Criteria:

1. Chronic or acute medical condition, including a history of seizures.
2. Body mass index 18-29.9 kg/m2
3. Current or previous major psychiatric disorder (e.g. psychotic disorders, mania / hypomania, anxiety disorders).
4. Psychotic or bipolar disorder in first-degree relatives, not including psychotic disorders secondary to an apparent medical reason, e.g., brain injury, dementia, or lesions of the brain.
5. Hypertension (SBP>140/90 mmHg) or hypotension (SBP<85 mmHg)
6. Psychedelic substance use (with the exception of cannabis) more than 20 times or any time within the previous two months
7. Pregnant or nursing women.
8. Participation in another clinical trial (currently or within the last 30 days).
9. Use of medications that may interfere with the effects of the study medications (any psychiatric medications and any medication with known to interact with the study substances).
10. Tobacco smoking (>10 cigarettes/day).
11. Consumption of alcoholic drinks (>15 drinks / week).
12. Body weight < 45 kg.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
5 dimensions of altered state of consciousness (5D-ASC) total OAV score | 10 hours after substance administration
  Visual analog scale consisting of 94 items. Constructed of five scales and allows assessing mood, anxiety, derealization, depersonalization, changes in perception, auditory alterations, and reduced vigilance. Scales will be presented as 100 mm long horizontal lines marked with vertical lines by the participant.

SECONDARY OUTCOMES:
Visual Analog Scales (VAS) good effect rating | One hour before, right after and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10 and 24 hours after substance administration
  VAS will be presented as 100 mm long horizontal lines marked with "not at all" on the left and "extremely" on the right. The following VAS items will be used: "any drug effect", "good drug effect", "bad drug effect", "drug high", "anxiety", "nausea", "feeling depressed", "alteration of vision", "alterations of hearing", "sounds seem to influence what I see", "alteration of sense of time", "the boundaries between myself and my surroundings seem to blur", "I gain insights into contexts that were previously were inscrutable to me", "talkative", "open", "trust" and "the context of my thought is personal/impersonal". Subjects will mark the scale with vertical lines.
Adjective Mood Rating Scale AMRS | One hour before as well as 3, 6, 10 and 24 hours after substance administration
  The adjective mood rating scale (AMRS or EWL60S) is a 60-item Likert scale that allows repeated assessment of mood in 6 dimensions: activation, inactivation, well-being, anxiety/depressed mood, extroversion and introversion, and emotional excitability.The AMRS consists of subscales measuring "activation", "positive mood", "extroversion", "introversion", "inactivation", and "emotional excitability.
States of consciousness questionnaire (SCQ) | 10 hours after substance administration
  This 100-item questionnaire is rated on a six-point scale. Forty-three items embedded into this questionnaire comprise the Mystical Experience Questionnaire (MEQ). which is sensitive to the effects of psilocybin. The 43 items provide scale scores for each of seven domains of mystical experiences: internal unity (pure awareness, a merging with ultimate reality), external unity (unity of all things, all things are alive, all is one), sense of sacredness (reverence, sacred), noetic quality (encounter with ultimate reality, more real than everyday reality), transcendence of time and space, deeply felt positive mood (joy, peace, love), paradoxicality/ineffability (claim of difficulty in describing the experience in words). The investigators will also derived the four scale scores of the newly validated revised 30-item MEQ: mystical, positive mood, transcendence of time and space, and ineffability.
Phenomenological-Autobiographical-Existential Psychedelic Scale extended (PAE-PS-ext) | This questionnaire is administrated once before the first substance day (during screening), and then again 10h after substance administration on everx study visit..
  This questionnaire rates psychedelic experiences with a focus on phenomenological, autobiographical, and existential psychedelic experiences. The scale includes 12 main questions to be answered on a total of 78 sub-ordered visual rating scales (sub-ordered visual rating scales mostly only need to be answered when the answer to the main question is "yes"). The last major question with eight sub-ordered visual rating scales of the PAE-PS is on worldview/beliefs.
Acute autonomic effects I (blood pressure) | One hour before, right after and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10 and 24 hours after substance administration
  Blood pressure (systolic and diastolic) will be measured with an automatic oscillometric device.
Acute autonomic effects II (heart rate) | One hour before, right after and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10 and 24 hours after substance administration
  Heart rate will be measured with an automatic oscillometric device.
Acute autonomic effects III (body temperature) | One hour before, right after and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10 and 24 hours after substance administration
  Body temperature will be measured with an ear thermometer.
Effect moderation by personality traits I (NEO-FFI) | Screening
  Personality traits are known to affect subjective responses to psychoactive substances and are assessed for explorative future analysis of pooled data. The NEO Five Factor Inventory (NEO-FFI) is a self-description questionnaire with 60 items for the measurement of the "big five": neuroticism, extraversion, openness, agreeableness, and consciousness. It uses a 5-point Likert scale ranging from "completely disagree" to "fully agree".
Effect moderation by personality traits II (FPI-R) | Screening
  Personality traits are known to affect subjective responses to psychoactive substances and are assessed for explorative future analysis of pooled data. The Freiburger Personality Inventory (FPI-R) version comprises 138 items and covers 12 dimensions of personality: life satisfaction, social orientation, performance orientation, inhibition, excitability, aggressiveness, stress, physical complaints, health concerns, openness, as well as the secondary factors according to Eysenck's Extraversion and Emotionality (Neuroticism). It uses a 2-point scale ("true" and "not true").
Effect moderation by personality traits III (SPF) | Screening
  Personality traits are known to affect subjective responses to psychoactive substances and are assessed for explorative future analysis of pooled data. The Saarbrücker Persönlichkeitsfragebogen (SPF) defines empathy as the "reactions of one individual to the observed experiences of another." It assesses 28-items on a 5-point Likert scale ranging from "Does not describe me well" to "Describes me very well". The measure has 4 subscales (Perspective Taking, Fantasy, Empathic Concern, Personal Distress) each made up of 7 different items.
Effect moderation by personality traits IV (HEXACO) | Screening
  Personality traits are known to affect subjective responses to psychoactive substances and are assessed for explorative future analysis of pooled data. The HEXACO personality inventory is a six-dimensional model of human personality with 100 items.The six factors are: Honesty-Humility, Emotionality, Extraversion, Agreeableness, Conscientiousness and Openness to Experience.
Effect moderation by personality traits V (DSQ-40) | Screening
  Personality traits are known to affect subjective responses to psychoactive substances and are assessed for explorative future analysis of pooled data. The Defense Style Questionnaire (DSQ-40) can provide scores for 20 individual defenses, and scores for the three factors "mature", "neurotic", and "immature". Each item is evaluated on a scale from 1 to 9, where "1" indicates "completely disagree" and "9" indicates "fully agree".
Psychological Insight Questionnaire (EBI+) | 10 hours after substance administration
  Assesses the degree of psychological insight caused by a psychedelic experience through 14-items to be answered on a 6-point Likert scale ranging from 0 ("not at all") to 5 ("extremely").
Changes in the electrocardiogram (ECG) | One hour before and 2 hours after substance administration.
  Corrected QT time (QTc) will be measured twice on the study days (baseline and at peak drug effect) to examine possible drug-induced changes in the ECG as well as a safety measure (millisecond scale).
Adverse effects (acute and subacute) | One hour before, 10 and 24 hours after substance administration
  The 2011 revised Beschwerden-Liste (B-LR) consists of a 40-item list covering a wide variety of symptoms and complaints that are answered with a four-point intensity-scoring ranging from "not at all" to "strong".
Persisting effects of the psychedelic experiences (PEQ) | End of study (EOS) visit during EOS interview
  140 items are rated on a six-point scale and include attitudes about life (13 positive and 13 negative items), attitudes about self (11 positive and 11 negative items), mood changes (nine positive and nine negative items), behavioral changes (one positive and one negative item), spirituality (22 positive and 21 negative items). Three additional questions are included
Cognitive Tasks | 24 hours after substance administration
  Cognitive assessment will be conducted using established tasks from the CANTAB battery. The tasks are administered in a computerized format.
Peak Plasma concentration of Psilocybin and Metabolites (Cmax) | Right after and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10 and 24 hours after substance administration
  Maximal Plasma concentration of Psilocybin and Metabolites Cmax after substance administration. Calculated via blood samples.
Time to cmax (Tmax) | Right after and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10 and 24 hours after substance administration
  Time until Psilocybin and Metabolites concentration peak in plasma after substance administration. Calculatet via blood samples after substance administration.
Area under the concentration-time curve up to 24 h (AUC0-24) | Right after and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10 and 24 hours after substance administration
  Area under the plasma concentration versus time curve for psilocybin and metaboliteswill be calculated up to 24h using blood sampels colected during the study visits after substance administration.
Elimination half life values (t1/2) | Right after and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10 and 24 hours after substance administration
  The elimination half life values of Psilocybin and metabolites will be calculated using blood samples collected during study visits after substance administration.
Sleep variables of %REM | 14 hours after substance administration until the end of the study day
  Sleep phases will be scored in every study session using an automated sleep stage classification algorithm of the SomnoArt® armband. The SomnoArt® armband will record, acceleration (3D accelerometer), and heart rate (red-infrared pulse oximeter) activity. Variables of %REM sleep is calculated as REM sleep duration divided by total sleep duration).
REM Latency | 14 hours after substance administration until the end of the study day
  Sleep phases will be scored in every study session using an automated sleep stage classification algorithm of the SomnoArt® armband. The SomnoArt® armband will record, acceleration (3D accelerometer), and heart rate (red-infrared pulse oximeter) activity. REM Latency is calculated as duration of non-REM sleep before the first REM phase.
REM Efficiency | 14 hours after substance administration until the end of the study day
  Sleep phases will be scored in every study session using an automated sleep stage classification algorithm of the SomnoArt® armband. The SomnoArt® armband will record, acceleration (3D accelerometer), and heart rate (red-infrared pulse oximeter) activity. REM Efficiency is calculated as REM sleep duration divided by the total REM episode duration

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Unit, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No